CLINICAL TRIAL: NCT00606268
Title: A Phase 1 Open-Label Study of the Safety and Pharmacokinetics of Repeated-Dose Micafungin as an Antifungal Prophylaxis in Children and Adolescents Undergoing Hematopoietic Stem Cell Transplant
Brief Title: A Study of Safety and Pharmacokinetics of Repeated Dose of Micafungin as Antifungal Prophylaxis in Children and Adolescents Who Undergo Hematopoietic Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9463-CL-2103
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Fungal Infections
Keywords: Antifungal Prophylaxis; Hematopoietic Stem Cell Transplant; HSCT; Micafungin
MeSH Terms: conditions — Mycoses | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 1.0 mg/kg
  Interventions: Drug: Micafungin
- 2 (Experimental): 1.5 mg/kg
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — IV
  Other Names: FK463

SUMMARY:
The study will evaluate PK and safety of two dose levels of Micafungin (FK463) as Antifungal prophylaxis in children and adolescents undergoing HSCT

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label, repeat-dose pharmacokinetic study that contains two treatment (micafungin 1.0mg/kg and 1.5mg/kg) dose groups. Subjects will be enrolled according to age and stratified by weight to receive either 1.0mg/kg (weight > 25kg) or 1.5mg/kg ( weight < 25kg) micafungin.

Children (4 months to < 2years, 2 to 5 years and 6 to 11 years) and adolescents (12 to 16 years) undergoing HSCT who require antifungal prophylaxis will be enrolled

ELIGIBILITY:
Inclusion Criteria:

* Institutional Review Board (IRB)-approved written informed Consent / Assent (as applicable) and HIPAA Authorization must be obtained from the subject (as able) and /or subject's parent/legally authorized representative prior to any study-related procedures
* Subject has sufficient venous access to permit administration of study drug, collect pharmacokinetic samples and monitor laboratory safety variables
* Female subject of childbearing potential must have a negative pregnancy test within 72 hours prior to the first dose of study drug, and if sexually active agree method of birth control per Investigator judgment for the duration of the study
* Subject (when able) and /or subjects parent/legally authorized representative agree to comply with the study requirements and with the concomitant medication restrictions
* Subject plans to undergo a HSCT

Exclusion Criteria:

* Subject has evidence of significant liver disease as defined by aspartate transamine (AST/SGOT), alanine transaminases (ALT/SGPT) 10 times the upper limit of normal (ULN) and total bilirubin or alkaline phosphatase > 5 times the ULN
* Subject has concomitant medical condition that in the opinion of the Investigator and /or medical monitor precludes enrollment into the study
* Subject with evidence of an active systemic or disseminated fungal infection prior to enrollment
* Subject has a history of anaphylaxis, hypersensitivity, or any serious reactions to the echinocandin class of antifungals
* Subject had received treatment with an echinocandin within one week prior to first dose of study drug
* Subject status is unstable and subject is unlikely to complete required study procedures
* Female subject is pregnant or nursing. Females of childbearing potential must avoid becoming pregnant while receiving study drug

Ages: 4 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Plasma drug concentration parameters: AUC0-24, Cmax | 13-17 Days

SECONDARY OUTCOMES:
Adverse events, vital signs, ECGs and laboratory test values | Day 1 to End of study

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Global Development
Locations (12):
- United States (12):
  - Los Angeles, California
  - Orange, California
  - Palo Alto, California
  - Denver, Colorado
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Minneapolis, Minnesota
  - Rochester, New York
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - Houston, Texas
  - Richmond, Virginia